CLINICAL TRIAL: NCT00882687
Title: A Phase 2, Single Center, Randomized, Double-Masked and Placebo Controlled Study Evaluating the Efficacy of Three Different Concentrations (0.1, 1.0, 5.0%) of SAR 1118 Ophthalmic Solution in a Modified Conjunctival Allergen Challenge (CAC) Model
Brief Title: Efficacy Study to Evaluate the Effectiveness of 3 Concentrations of SAR 1118 in Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1118-ACJ-100
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.1% Lifitegrast (Experimental)
  Interventions: Drug: Lifitegrast
- 1.0% Lifitegrast (Experimental)
  Interventions: Drug: Lifitegrast
- 5.0% Lifitegrast (Experimental)
  Interventions: Drug: Lifitegrast
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lifitegrast — Ophthalmic Solution
  Other Names: SAR 1118
  Arms: 0.1% Lifitegrast; 1.0% Lifitegrast; 5.0% Lifitegrast
Other: Placebo — Ophthalmic Solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether SAR 1118 at three different concentrations, compared to placebo, is effective in the prevention of the signs and symptoms of allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form and HIPAA document
* Willing and able to comply with all study procedures
* Be at least 18 years of age at the time of enrollment
* 20/40 vision, or better, in each eye
* History of ocular allergies, and a positive skin and ocular allergic reaction to allergens
* A negative urine pregnancy test if female of childbearing potential and must use adequate birth control throughout the study period

Exclusion Criteria:

* Preauricular lymphadenopathy or any ocular condition that could affect study parameters (particularly, glaucoma, diabetic retinopathy, clinically significant blepharitis, follicular conjunctivitis and iritis)
* Have had any ocular infection within the last 30 days
* A positive diagnosis of moderate to severe dry eye syndrome (i.e., requiring daily use of artificial tears)
* Any significant illness that could be expected to interfere with study parameters
* Manifest signs or symptoms of clinically active allergic conjunctivitis in either eye
* Use of any investigational product or device within one month prior to Visit 1 or during the study period
* Concomitant use of any prohibited medication (antihistamines, corticosteroids, all ocular medications or anti-allergic therapies) during the trial or within the washout period
* Any blood donation or significant loss of blood within 56 days of Visit 1
* Any history of autoimmune disease, immunodeficiency disorder, positive HIV, hepatitis B, C, or evidence of acute active hepatitis A (anti-HAV IgM), or organ or bone marrow transplant. Any known history of iritis/uveitis, glaucoma, or other chronic ophthalmologic disorder other than allergic conjunctivitis
* History of laser-assisted in situ keratomileusis (LASIK) or similar type of corneal refractive surgery within 12 months prior to Visit 1, and/or any other ocular surgical procedure within 3 months prior to Visit 1
* Known history of alcohol abuse and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04-24 (Actual); Primary Completion 2009-05-10 (Actual); Study Completion 2009-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Ora, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Started | 15 | 15 | 15 | 15
Completed | 13 | 13 | 12 | 13
Not Completed | 2 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included data from all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.67 (15.207) | 37.67 (12.613) | 45.33 (15.891) | 39.13 (12.212) | 40.95 (14.019)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 9 | 6 | 29
  Male | 6 | 10 | 6 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching at Day 7 (7 Minutes Post Conjunctival Allergen Challenge [CAC 6])
Description: Ocular Itching was evaluated by participants and graded with Ophthalmic Research Associates, Inc. (ORA) Scale with the score ranged from 0 to 4 (0=none; 0.5=intermittent tickle in the cornea; 1=intermittent tickle more than just the cornea; 1.5=intermittent all-over tickling sensation; 2=mild conscious itch without desire to rub; 2.5=moderate, diffuse continuous itch with desire to rub; 3=severe itch with desire to rub; 3.5=severe itch improved with minimal rubbing; 4=incapacitating itch with an irresistible urge to rub) with 0.5 point increments allowed, and lower scores indicates lesser ocular itching. CAC is an initial titration challenge to determine the appropriate allergen and lowest concentration of allergen that produced a positive bilateral allergic response for each subject, defined as ≥ 2 score (0-4 point scale) in ocular itching and conjunctival redness within 10 minutes of the last titration of allergen.
Time Frame: Baseline to Day 7 (7 minutes post CAC 6)
Population: Intent-to-treat (ITT) population with last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 2.65 (0.731) | 2.68 (1.096) | 3.07 (0.837) | 2.88 (0.410)
Statistical Analysis 1: Comparison: Lifitegrast 0.1% vs Placebo; Test type: Superiority or Other; p = 0.3235, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Lifitegrast 1.0% vs Placebo; Test type: Superiority or Other; p = 0.9144, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Lifitegrast 5.0% vs Placebo; Test type: Superiority or Other; p = 0.3324, Wilcoxon rank-sum test

2. Primary Outcome: Ocular Itching at Day 14 (7 Minutes Post CAC 9)
Description: Ocular Itching was evaluated by participants and graded with Ophthalmic Research Associates, Inc. (ORA) Scale with the score ranged from 0 to 4 (0=none; 0.5=intermittent tickle in the cornea; 1=intermittent tickle more than just the cornea; 1.5=intermittent all-over tickling sensation; 2=mild conscious itch without desire to rub; 2.5=moderate, diffuse continuous itch with desire to rub; 3=severe itch with desire to rub; 3.5=severe itch improved with minimal rubbing; 4=incapacitating itch with an irresistible urge to rub) with 0.5 point increments allowed, and lower scores indicates lesser ocular itching.
Time Frame: Baseline to Day 14 (7 minutes post CAC 9)
Population: ITT population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 2.28 (1.043) | 2.50 (1.191) | 2.63 (0.968) | 2.12 (0.737)
Statistical Analysis 1: Comparison: Lifitegrast 0.1% vs Placebo; Test type: Superiority or Other; p = 0.5846, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Lifitegrast 1.0% vs Placebo; Test type: Superiority or Other; p = 0.1493, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Lifitegrast 5.0% vs Placebo; Test type: Superiority or Other; p = 0.0404, Wilcoxon rank-sum test

3. Primary Outcome: Conjunctival Redness at Day 7 (20 Minutes Post CAC 6)
Description: Conjunctival Redness was evaluated by an investigator with slit lamp and graded with ORA Scale with the score ranged from 0 to 4 (0=none; 1=mild-slightly dilated blood vessels; color of vessels is typically pink; can be quadrantal; 2=moderate-more apparent dilation of blood vessels; vessel color is more intense (redder); involves the majority of the vessel bed; 3=severe-numerous and obvious dilated blood vessels; in the absence of chemosis the color is deep red, may be less red or pink in presence of chemosis, is not quadrantic; 4=extremely severe-large, numerous, dilated blood vessels characterized by unusually severe deep red color, regardless of grade of chemosis, which involves the entire vessel bed) with 0.5 point increments allowed, and lower scores indicates reduction in the conjunctival redness.
Time Frame: Baseline to Day 7 (20 minutes post CAC 6)
Population: ITT population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 2.27 (0.458) | 2.48 (0.406) | 2.57 (0.477) | 2.52 (0.427)
Statistical Analysis 1: Comparison: Lifitegrast 0.1% vs Placebo; Test type: Superiority or Other; p = 0.0578, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Lifitegrast 1.0% vs Placebo; Test type: Superiority or Other; p = 0.8988, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Lifitegrast 5.0% vs Placebo; Test type: Superiority or Other; p = 0.4709, Wilcoxon rank-sum test

4. Primary Outcome: Conjunctival Redness at Day 14 (20 Minutes Post CAC 9)
Description: as for outcome 3
Time Frame: Baseline to Day 14 (20 minutes post CAC 9)
Population: ITT population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale | 1.92 (0.686) | 2.42 (0.397) | 2.38 (0.399) | 2.17 (0.652)
Statistical Analysis 1: Comparison: Lifitegrast 0.1% vs Placebo; Test type: Superiority or Other; p = 0.1773, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Lifitegrast 1.0% vs Placebo; Test type: Superiority or Other; p = 0.4222, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Lifitegrast 5.0% vs Placebo; Test type: Superiority or Other; p = 0.4326, Wilcoxon rank-sum test

5. Secondary Outcome: Ocular Itching at Day 6 (CAC 4), 5 (CAC 7)
Description: as for outcome 2
Time Frame: Baseline to Day 6 (CAC 4), Day 13 (CAC 7) 7 minutes post CAC
Population: ITT population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale
  Visit 3: 7 minutes post CAC 4 | 2.83 (0.564) | 2.37 (0.886) | 3.02 (0.644) | 2.82 (0.395)
  Visit 5: 7 minutes post CAC 7 | 2.42 (1.084) | 2.62 (0.778) | 2.63 (0.972) | 2.38 (0.388)

6. Secondary Outcome: Conjunctival Redness at Day 6 (CAC 4), 5 (CAC 7)
Description: as for outcome 3
Time Frame: Baseline to Day 6 (CAC 4), Day 13 (CAC 7) at 20 minutes post CAC
Population: ITT population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
units on a scale
  Visit 3: 20 minutes post CAC 4 | 1.82 (0.594) | 2.15 (0.725) | 2.25 (0.605) | 2.25 (0.433)
  Visit 5: 20 minutes post CAC 7 | 1.37 (0.911) | 2.15 (0.749) | 1.62 (1.026) | 1.77 (0.863)

ADVERSE EVENTS:
Time Frame: Up to Day 16
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 6/15 | 7/15 | 12/15 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast 0.1% (N=15) | Lifitegrast 1.0% (N=15) | Lifitegrast 5.0% (N=15) | Placebo (N=15)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast 0.1% (N=15) | Lifitegrast 1.0% (N=15) | Lifitegrast 5.0% (N=15) | Placebo (N=15)
Eye Disorders (Eye disorders) | 4 (7) | 6 (11) | 9 (16) | 0 (0)
General Discomfort and Administration Site Conditions (General disorders) | 4 (5) | 2 (3) | 6 (10) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.